CLINICAL TRIAL: NCT04991571
Title: A Phase 1, Open-label Study With Two Independent Parts: Collecting Samples for Metabolites in Safety Testing Analysis of Zibotentan After Repeated Administration (Part 1); and a Randomised, Cross-over, Three Period, Three-treatment, Single Dose Study to Assess the Relative Bioavailability of Different Formulations of Zibotentan and Dapagliflozin (Part 2) in Healthy Adult Participants
Brief Title: Study to Collect Samples for MIST Analysis of Zibotentan and Bioavailability of Zibotentan and Dapagliflozin in Heatlhy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D4325C00003
Record Dates: First submitted 2021-07-28; First posted 2021-08-05 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — ZD4054; dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1 (Experimental): Participants will be administered with zibotentan once daily for 5 days.
  Interventions: Drug: Zibotentan (Treatment A)
- Part 2: Treatment Sequence ABC (Experimental): Each participant will receive 3 single-dose treatments of zibotentan and dapagliflozin (Treatment A; Treatment B; Treatment C) in 3 treatment periods, separated by a washout period of at least 7 days between treatment periods.
  Interventions: Drug: Zibotentan (Treatment A); Drug: Dapagliflozin (Treatment A); Drug: Zibotentan/Dapagliflozin - Formulation 1 (Treatment B); Drug: Zibotentan/Dapagliflozin - Formulation 2 (Treatment C)
- Part 2: Treatment Sequence BCA (Experimental): Each participant will receive 3 single-dose treatments of zibotentan and dapagliflozin (Treatment B; Treatment C; Treatment A) in 3 treatment periods, separated by a washout period of at least 7 days between treatment periods.
  Interventions: Drug: Zibotentan (Treatment A); Drug: Dapagliflozin (Treatment A); Drug: Zibotentan/Dapagliflozin - Formulation 1 (Treatment B); Drug: Zibotentan/Dapagliflozin - Formulation 2 (Treatment C)
- Part 2: Treatment Sequence CAB (Experimental): Each participant will receive 3 single-dose treatments of zibotentan and dapagliflozin (Treatment C; Treatment A; Treatment B) in 3 treatment periods, separated by a washout period of at least 7 days between treatment periods.
  Interventions: Drug: Zibotentan (Treatment A); Drug: Dapagliflozin (Treatment A); Drug: Zibotentan/Dapagliflozin - Formulation 1 (Treatment B); Drug: Zibotentan/Dapagliflozin - Formulation 2 (Treatment C)

INTERVENTIONS:
Drug: Zibotentan (Treatment A) — Zibotentan capsule will be administered orally as multiple doses in Part 1 and as single dose in Part 2.
Drug: Dapagliflozin (Treatment A) — Dapagliflozin tablet will be administered orally as single dose in Part 2.
  Arms: Part 2: Treatment Sequence ABC; Part 2: Treatment Sequence BCA; Part 2: Treatment Sequence CAB
Drug: Zibotentan/Dapagliflozin - Formulation 1 (Treatment B) — Zibotentan/Dapagliflozin tablet will be administered orally as single dose in Part 2.
  Arms: Part 2: Treatment Sequence ABC; Part 2: Treatment Sequence BCA; Part 2: Treatment Sequence CAB
Drug: Zibotentan/Dapagliflozin - Formulation 2 (Treatment C) — Zibotentan/Dapagliflozin tablet will be administered orally as single dose in Part 2.
  Arms: Part 2: Treatment Sequence ABC; Part 2: Treatment Sequence BCA; Part 2: Treatment Sequence CAB

SUMMARY:
The study will have 2 independent parts:

Part 1 of the study is intended to collect samples for Metabolites in Safety Testing (MIST) analysis after administration of multiple doses of zibotentan.

Part 2 of the study is designed to evaluate the relative bioavailability of zibotentan and dapagliflozin after dosing with two different fixed-dose combination (FDC) formulations and dosing with separate formulations of zibotentan and dapagliflozin.

DETAILED DESCRIPTION:
Part 1 will be an open-label, non-randomised, single treatment period. A single treatment period during which participants will be resident at the study centre from 2 days before dosing (Day -2) until the morning of Day 6.

Part 2 will be an open-label, randomised, 3-period, 3-treatment, cross-over single dose study. Participants will be randomised to one of 3 treatment sequences and will receive 3 single-dose study interventions. Participants will be resident at the study centre from 2 days before dosing (Day -2) until Day 3 of the last treatment sequence.

Participants who were enrolled in Part 1 may not be enrolled in Part 2.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study participants should fulfil the following criteria:

1. Participants with suitable veins for cannulation or repeated venipuncture.
2. Females must have a negative pregnancy test at the Screening Visit and within 24 hours prior to dosing, must not be lactating and must be of non- childbearing potential
3. Male participant must adhere to the contraception methods.
4. Have a BMI between 18 and 29.9 kg/m^2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.
5. Provision of signed and dated, written informed consent prior to any study specific procedures.

Exclusion Criteria:

Participants will not enter the study if any of the following exclusion criteria are fulfilled:

1. History or presence of gastrointestinal, hepatic or renal disease or any important disease or disorder.
2. Any clinically important illness, medical/surgical procedure or trauma within 4 weeks of the first administration of study intervention.
3. Any clinically significant abnormalities in clinical chemistry, haematology, or urinalysis.
4. Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody, and Human immunodeficiency virus antibody.
5. Abnormal vital signs. 6 History of drug abuse or alcohol abuse.

7. History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity.

8. Participants who are vegans or have medical dietary restrictions. 9. Participants tested positive for COVID-19 at the time of randomisation or have been previously hospitalised with COVID-19 infection.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2021-10-22 (Actual); Study Completion 2021-10-22 (Actual)

PRIMARY OUTCOMES:
Part 1: Metabolites in Safety Testing sampling | Day 1 through Day 6 (pre-dose, 30 min; 1, 2, 4, 6, 8, 12 and 24 hours post dose)
  Plasma sample will be collected to understand the PK profiling of zibotentan metabolites and to meet the regulatory requirements.
Part 2: Area under plasma concentration time curve from zero to infinity (AUCinf) | Day 1 through Day 3 of each treatment period
  Relative bioavailability of zibotentan and dapagliflozin after dosing with two different FDC formulations and dosing with separate formulations of zibotentan and dapagliflozin will be evaluated.
Part 2: Area under the plasma concentration curve from zero to the last quantifiable concentration (AUClast) | Day 1 through Day 3 of each treatment period
  Relative bioavailability of zibotentan and dapagliflozin after dosing with two different FDC formulations and dosing with separate formulations of zibotentan and dapagliflozin will be evaluated.
Part 2: Maximum observed plasma drug concentration (Cmax) | Day 1 through Day 3 of each treatment period
  Relative bioavailability of zibotentan and dapagliflozin after dosing with two different FDC formulations and dosing with separate formulations of zibotentan and dapagliflozin will be evaluated.
Part 2: Observed concentration at 24 hours post-dose (C24) | Day 1 through Day 3 of each treatment period
  Relative bioavailability of zibotentan and dapagliflozin after dosing with two different FDC formulations and dosing with separate formulations of zibotentan and dapagliflozin will be evaluated.

SECONDARY OUTCOMES:
Part 2: Time to reach peak or maximum observed concentration (tmax) | Day 1 through Day 3 of each treatment period
  Relative bioavailability of zibotentan and dapagliflozin after dosing with two different FDC formulations and dosing with separate formulations of zibotentan and dapagliflozin will be evaluated.
Part 2: Terminal rate constant (λz) | Day 1 through Day 3 of each treatment period
  Relative bioavailability of zibotentan and dapagliflozin after dosing with two different FDC formulations and dosing with separate formulations of zibotentan and dapagliflozin will be evaluated.
Part 2: Half life associated with λz (t½λz) | Day 1 through Day 3 of each treatment period
  Relative bioavailability of zibotentan and dapagliflozin after dosing with two different FDC formulations and dosing with separate formulations of zibotentan and dapagliflozin will be evaluated.
Part 2: Apparent total body clearance of drug from plasma after extravascular administration (CL/F) | Day 1 through Day 3 of each treatment period
  Relative bioavailability of zibotentan and dapagliflozin after dosing with two different FDC formulations and dosing with separate formulations of zibotentan and dapagliflozin will be evaluated.
Part 2: Volume of distribution at steady state following extravascular administration (Vz/F) | Day 1 through Day 3 of each treatment period
  Relative bioavailability of zibotentan and dapagliflozin after dosing with two different FDC formulations and dosing with separate formulations of zibotentan and dapagliflozin will be evaluated.
Part 1 and Part 2: Number of adverse events and serious adverse events | From Sceerning to Follow-up Visit approximately 40 days for Part 1 and 49 days for Part 2
  Safety and tolerability of zibotentan and dapagliflozin will be studied.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Brooklyn, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home